CLINICAL TRIAL: NCT06977919
Title: Efficacy of a 12-Week NASM Optimum Performance Training Program on Pectoral Muscle Strength, Breast Aesthetics, and Low Back Pain in Non-Athletic Women: A Randomized Controlled Trial
Brief Title: NASM OPT for Pectoral Enhancement and Breast Firmness in Non-Athletic Women: An RCT
Acronym: BreastFirmne
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sistan and Baluchestan (Other)
Responsible Party: Principal Investigator, Mohammadreza Rezaeipour, Assoc.Prof.Dr., University of Sistan and Baluchestan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 9378-30-3-2025
Record Dates: First submitted 2025-05-10; First posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Low Back Pain; Muscle Weakness; Breast Sagging
Keywords: NASM OPT; Pectoral Muscles; Breast Firmness; Non-Athletic Women; Resistance Training
MeSH Terms: conditions — Low Back Pain; Muscle Weakness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Single-blind (outcome assessors only; participants/instructors unblinded due to intervention nature).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NASM OPT Group (Experimental): Three 60-minute weekly sessions for 12 weeks, progressing through stabilization (weeks 1-4), strength endurance (weeks 5-8), and hypertrophy (weeks 9-12) phases. Exercises included bench presses, chest flyes, and push-ups.
  Interventions: Behavioral: NASM OPT Program
- General Exercise Group (Active Comparator): Three 60-minute weekly sessions of brisk walking and light aerobics without targeted resistance training.
  Interventions: Behavioral: General Exercise

INTERVENTIONS:
Behavioral: NASM OPT Program — Three 60-minute weekly sessions for 12 weeks, progressing through stabilization (weeks 1-4), strength endurance (weeks 5-8), and hypertrophy (weeks 9-12) phases. Exercises included bench presses, chest flyes, and push-ups.
  Other Names: Experimental
  Arms: NASM OPT Group
Behavioral: General Exercise — Three 60-minute weekly sessions of brisk walking and light aerobics without targeted resistance training.
  Other Names: Active Comparator
  Arms: General Exercise Group

SUMMARY:
This RCT investigates a 12-week NASM OPT program targeting pectoral muscle strength, breast aesthetics (firmness, lift, chest circumference), and low back pain in 120 non-athletic women. The intervention group performed structured resistance training, while the control group engaged in general exercise. Outcomes included pectoral strength (dynamometer), aesthetic satisfaction (Likert scale), and functional performance (push-up test).

DETAILED DESCRIPTION:
Participants were randomized to NASM OPT (3 weekly sessions: stabilization, strength, and hypertrophy phases) or general exercise (brisk walking/aerobics). Measurements at baseline and 12 weeks included pectoral strength, chest circumference, low back pain (VAS), and perceived breast aesthetics.

ELIGIBILITY:
Inclusion Criteria:

* Non-athletic women (no exercise in prior 6 months).
* Interest in improving chest aesthetics.
* No musculoskeletal injuries.

Exclusion Criteria:

* Pregnancy
* Chronic illness
* Exercise contraindications

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 120 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-08-15 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Pectoral Strength | Baseline, 12 weeks
  Kilogram (kg); handheld dynamometer
Perceived Breast Firmness/Lift | Baseline, 12 weeks
  5-point Likert scale
Chest Circumference | Baseline, 12 weeks
  Centimeter (cm)

SECONDARY OUTCOMES:
Aesthetic Satisfaction | Baseline, 12 weeks (post-intervention)
  5-point Likert scale
Functional Performance | Baseline, 12 weeks (post-intervention)
  30-second push-up test
Low Back Pain | Baseline, 12 weeks (post-intervention)
  VAS, 0-10 cm

CONTACTS AND LOCATIONS:
Overall Officials: Mohammadreza Rezaeipour, MD, PhD, Study Director — Assoc.Prof.Dr.
Locations (1):
- Sport Sciences Department, Zahedan, Sistan and Baluchestan, Iran

IPD SHARING:
Plan to Share IPD: No
Privacy concerns regarding sensitive participant data.